CLINICAL TRIAL: NCT06190145
Title: A Single-arm, Open-label Phase II Study to Determine the Safety and Efficacy of Teriflunomide in Patients With Steroid-resistant/Relapse Thrombocytopenia
Brief Title: Teriflunomide for Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-TFITP-02
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Immune Thrombocytopenia
Keywords: Teriflunomide
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teriflunomide (Experimental): Oral Teriflunomide is given at a dose of 7 mg once daily with dose adjustments for 24 weeks. Treatment was discontinued if a dose-limiting toxic effect occurred, rescue medication was used, or concomitant medication for immune thrombocytopenia was changed beyond the 10% level as defined above.
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Starting dose of 7 mg once daily. Dose adjustments were made throughout the study based on individual platelet counts.
  Other Names: AUBAGIO

SUMMARY:
Single-arm, open-label, single-center study to evaluate the efficacy and safety of teriflunomide for the treatment of adults with steroid-resistant/relapse immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label study of teriflunomide in approximately 40 patients with ITP who have relapsed or have an insufficient response to prior therapies. Teriflunomide is administered as 7 mg orally once daily with dose adjustments for 24 weeks. Efficacy and safety outcomes are assessed on scheduled study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary immune thrombocytopenia (ITP) by excluding other supervened causes of thrombocytopenia
2. Patients with a platelet count <30,000/μL or a platelet count <50,000/μL with bleeding manifestations at the enrollment;
3. Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid tapering or after its discontinuation;
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Secondary immune thrombocytopenia (e.g. patients with HIV, HCV, Helicobacter pylori infection, malignancy, or patients with confirmed autoimmune disease);
3. Pregnancy or lactation;
4. Pre-existing acute or chronic liver disease, or serum alanine aminotransferase (ALT) greater than 2 times the upper limit of normal (ULN);
5. Current or recent (< 4 weeks prior to screening) clinically serious viral, bacterial, fungal, or parasitic infection;
6. Have evidence of active tuberculosis (TB), or have previously had evidence of active TB and did not receive appropriate and documented treatment, or have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB;
7. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Sustained response | From the start of study treatment (Day 1) to the end of week 24
  Platelet count over 30,000/μL and at least a 2-fold increase of the baseline count in the absence of bleeding and rescue therapy for at least four of the six visits between weeks 19 and 24.

SECONDARY OUTCOMES:
Overall response | From the start of study treatment (Day 1) to the end of week 24
  Complete response (CR) was defined as platelet count over 100,000/μL and absence of bleeding. Response (R) was defined as platelet count over 30,000/μL and at least a 2-fold increase of the baseline count and absence of bleeding.
Initial response | From the start of study treatment (Day 1) up to week 4 of treatment
  The number of participants with achievement of CR or R at 4 weeks.
Time to response | From the start of study treatment (Day 1) to the end of week 24
  The time from treatment initiation to achieve a CR or a R.
Bleeding events | From the start of study treatment (Day 1) to the end of week 24
  Clinically significant bleeding was assessed using the World Health Organization (WHO) bleeding scale.
Adverse events | From the start of study treatment (Day 1) to the end of week 24
  Adverse events (AEs) were reported and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) to the end of week 24
  ITP-PAQ was used to assess the Health-Related Quality of Life (HRQoL) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, China